CLINICAL TRIAL: NCT00370201
Title: Efficacy of Oral Colchicine in Prevention of Proliferative Vitreoretinopathy in Rhegmatogenous Retinal Detachment
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Shahid Beheshti University of Medical Sciences (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 8259
Record Dates: First submitted 2006-08-30; First posted 2006-08-31 (Estimated); Last update posted 2006-10-09 (Estimated); Status verified 2004-03

CONDITIONS: Rhegmatogenous Retinal Detachment
Keywords: retinal detachment; proliferative vitreoretinopathy
MeSH Terms: conditions — Retinal Detachment; Vitreoretinopathy, Proliferative | interventions — Colchicine

INTERVENTIONS:
Drug: colchicine

SUMMARY:
This clinical trial will test the efficacy and safety of oral colchicine in prevention of proliferative vitreoretinopathy (PVR) in cases of rhegmatogenous retinal detachment

ELIGIBILITY:
Inclusion Criteria:

* Rhegmatogenous retinal detachment

Exclusion Criteria:

* PVR grade C
* Duration of retinal detachment ≥ one month
* History of cataract surgery
* History of RD surgery

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2004-03; Study Completion 2006-08

PRIMARY OUTCOMES:
proliferative vitreoretinopathy
retinal reattachment rate

SECONDARY OUTCOMES:
visual acuity
reoperation
macular pucker

CONTACTS AND LOCATIONS:
Overall Officials: Hamid Ahmadieh, MD, Principal Investigator — Ophthalmic Research Center of Shaheed Beheshti Medical University
Locations (1):
- Hamid Ahmadieh,MD, Tehran, Tehran Province, Iran